CLINICAL TRIAL: NCT05655793
Title: The TearAD Study: Tear Biomarkers for Alzheimer's Disease (AD) Screening and Diagnosis
Acronym: TearAD
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-033
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: Tear Fluid; Retinal imaging; Biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The type of biospecimen that is retained is tear fluid collected with Schirmer's strips, CSF and blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Neurodegeneration: Includes patients with mild cognitive impairment and dementia
  Interventions: Diagnostic Test: Tear Fluid collection (Schirmer's strip); Diagnostic Test: Retinal imaging
- Without Neurodegeneration: Includes healthy controls and patients with subjective cognitive decline
  Interventions: Diagnostic Test: Tear Fluid collection (Schirmer's strip); Diagnostic Test: Retinal imaging

INTERVENTIONS:
Diagnostic Test: Tear Fluid collection (Schirmer's strip) — Tear fluid will be collected non-invasively form all participants with the use of Schirmer's strips, which is a small paper strip placed in the lower eye lid for a maximum of 5 minutes.
Diagnostic Test: Retinal imaging — The retina from all participants will be visualised with the use of a standard (Clarus 700 Zeiss), ultra-wide field (Optos), and cross-sectional (Optical Coherence Tomography) retinal images.

SUMMARY:
The goal of this observational longitudinal study is to investigates whether tear fluid is a non-invasive source of biomarkers for Alzheimer's disease. The main aim of the study is to evaluate diagnostic accuracy measures (sensitivity and specificity) of tear and retinal biomarkers to discriminate individuals with and without neurodegeneration.

Tear fluid from participants will be collected non-invasively with Schirmer's strips, which is a small paper strip placed in the lower eye lid for a maximum of 5 minutes. Additionally, standard, ultra-wide field and cross-sectional retinal images will be obtained.

ELIGIBILITY:
Inclusion Criteria (healthy controls):

* Available CSF, PET, CT or MRI data to evaluate the presence/absence of neurodegeneration (preferably within 1 year of inclusion in this study)
* Absence of cognitive complaints or treatment and did not seek help for cognitive complaints in the past
* MMSE score 26-30 at baseline
* Age > 50 years
* Available for follow-up (up to 24 months)
* Written informed consent obtained and documented

Inclusion criteria (patients):

* Available CSF, PET, CT or MRI data to evaluate the presence/absence of neurodegeneration (preferably within 1 year of inclusion in this study)
* Available for follow-up (up to 24 months)
* Written informed consent obtained and documented
* Capable of giving informed consent themselves (MMSE score > 17/30)

Exclusion Criteria (all subjects):

* Ocular conditions that could influence tear biochemical parameters (including eye infection, eye inflammation, eye surgery within the last 28 days or other acute eye conditions)
* Neurological or systemic chronic conditions known to interfere with retinal thickness (e.g., glaucoma, diabetes mellitus)
* Ocular conditions interfering with optical coherence tomography (OCT) quality/retinal thickness: e.g. severe cataract, age-related macular degeneration, and glaucoma

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from the population that visit the memory clinic and are willing to participate in scientific research.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Capability of tear biomarkers to discriminate individuals with neurodegeneration from those without neurodegeneration and assess the change in biomarker levels over time. | Sampling done at t= 0, 1 and 2 years.
  Levels of tear biomarkers will be determined from the Schirmer's strips. The biomarker levels will be analysed to see whether they can be discriminate between people with and without neurodegeneration.

SECONDARY OUTCOMES:
The difference in tear biomarker level between patients and controls, and between patient groups and how these differences change over time. | Sampling done at t= 0, 1 and 2 years.
  Additional analysis to see whether tear biomarkers can also discriminate patients from controls and differences inbetween patient groups.
Correlation of biomarker levels in tears, blood and cerebral spinal fluid (CSF). | Baseline measurements (t=0) will be used to determine correlation.
  This analysis will be done to determine the correlation between biomarkers of different body fluids.
Correlation between tear biomarkers and other ocular imaging biomarkers, as well as assessing the change of this correlation over time. | Imaging done at t= 0, 1 and 2 years.
  The correlation between tear biomarkers and ocular imaging biomarkers (e.g. thickness of the retinal nerve fiber layer, retinal vasculature tortuosity) will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Gijs, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Academic Hospital Maastricht, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van de Sande N, Ramakers IHGB, Visser PJ, Verhey FRJ, Verbraak FD, Bouwman FH, Berendschot TTJM, Nuijts RMMA, Webers CAB, Gijs M. Tear biomarkers for Alzheimer's disease screening and diagnosis (the TearAD study): design and rationale of an observational longitudinal multicenter study. BMC Neurol. 2023 Aug 5;23(1):293. doi: 10.1186/s12883-023-03335-y. PMID 37543602